CLINICAL TRIAL: NCT02682563
Title: A Randomized, Double-blind, Comparator-controlled Trial to Assess the Effect of 12-week Treatment With Dapagliflozin Versus Gliclazide on Renal Physiology and Biomarkers in Metformin-treated Patients With Type 2 Diabetes Mellitus
Brief Title: Renoprotective Effects of Dapagliflozin in Type 2 Diabetes
Acronym: RED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.H.H. Kramer (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, M.H.H. Kramer, Head of the Internal Medicine department, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DC 2015 RED 01; 2015-003818-24 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-15 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathies
Keywords: SGLT-2 inhibition, Renal, Cardiovascular, Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — dapagliflozin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin 10mg once daily (Experimental): Once daily treatment with oral dapagliflozin (forxiga) 10mg for 12 consecutive weeks.
  Interventions: Drug: Dapagliflozin 10mg QD
- Gliclazide modified release 30mg once daily (Active Comparator): Once daily treatment with oral gliclazide MR 30mg for 12 consecutive weeks.
  Interventions: Drug: Gliclazide 30mg QD

INTERVENTIONS:
Drug: Dapagliflozin 10mg QD — Dapagliflozin 10mg once daily for 12 weeks
  Other Names: forxiga
  Arms: Dapagliflozin 10mg once daily
Drug: Gliclazide 30mg QD — Gliclazide30mg once daily for 12 weeks
  Other Names: Diamicron
  Arms: Gliclazide modified release 30mg once daily

SUMMARY:
Background:

Worldwide, diabetic nephropathy or Diabetic Kidney Disease (DKD), is the most common cause of chronic and end-stage kidney disease. With the increasing rates of obesity and type 2 diabetes (T2DM), many more patients with DKD may be expected in the coming years. Large-sized prospective randomized clinical trials suggest that intensified glucose and blood pressure control, may halt the progression of DKD, both in type 1 diabetes and T2DM. However, despite the wide use of angiotensin-converting enzyme inhibitors and angiotensin receptor blockers, a considerable amount of patients develop DKD during the course of diabetes, indicating an unmet need for renoprotective therapies. Sodium-glucose linked transporters (SGLT-2) inhibitors are novel glucose-lowering drugs for the treatment of T2DM. These agents seem to exert pleiotropic actions 'beyond glucose control', including reduction of blood pressure and body weight. In addition, SGLT-2 inhibitors decrease proximal sodium reabsorption and decrease glomerular pressure and albuminuria in rodents and type 1 diabetes patients. In rodents, SGLT-2 inhibitors also improved histopathological abnormalities associated with DKD. To date, the potential renoprotective effects and mechanisms of these agents have not been sufficiently detailed in human type 2 diabetes. The current study aims to explore the clinical effects and mechanistics of SGLT-2 inhibitors on renal physiology and biomarkers in metformin-treated T2DM patients with normal kidney function.

Study Design:

Randomized, double-blind, comparator-controlled, intervention trial

Study Endpoints:

Renal hemodynamics, i.e. measured glomerular filtration rate (GFR, ml/min) and effective renal plasma flow (ERPF, ml/min); 24-hour urinary solute excretion; markers of renal damage ; blood pressure; body anthropometrics; systemic hemodynamic variables (including stroke volume, cardiac output and total peripheral resistance); arterial stiffness will be assessed by applanation tonometry, (SphygmoCor®); insulin sensitivity and beta-cell function.

Expected results:

Treatment with the SGLT-2 inhibitor dapagliflozin, as compared to the sulfonylurea (SU) derivative gliclazide, may confer renoprotection by improving renal hemodynamics, and decreasing blood pressure and body weight in type 2 diabetes.

DETAILED DESCRIPTION:
Study design A phase 4, monocenter, randomized, double-blind, comparator-controlled, parallel-group, mechanistic intervention trial to assess the effect of 12-week treatment with the sodium-glucose linked transporters (SGLT)-2 inhibitor dapagliflozin versus the sulfonylurea (SU) derivative gliclazide on renal physiology and biomarkers in metformin-treated patients with type 2 diabetes mellitus (T2DM)

Recruitment Subjects will be recruited by researcher physicians involved in this trial using methods that are established practice for all human studies in the Diabetes Center, Vrije Universiteit (VU) University Medical Center (VUMC), via advertisements, use of a Diabetes Center database, through the Diabetes Center website.

Screening and eligibility After giving extensive oral and written information, a written informed consent form will be obtained from the subjects before screening. The screening procedure will consist of obtaining an extensive medical history, complete physical examination, blood analysis, urine screening, and a 12-lead electrocardiogram (ECG). Postvoid residual urine volume will be determined by ultrasonic bladder scan. After inclusion, participants will enroll in a 4-week run-in period to allow for study effects.

Baseline assessments Seven days prior to this visit, subjects will adhere to a 'normal-salt' (9 - 12 grams or 150 - 200 mmol per day) and protein (1.5 - 2.0 g/kg per day) diets, in order to minimize variation in renal physiology due to salt and protein intake. Participants will abstain from alcohol (24 hours), caffeine (12 hours) and nicotine (12 hours) and heavy exercise prior to and during visits 2. One day prior to the testing day, subjects will collect 24-hour urine.

Following an overnight fast, participants will be instructed to drink 500 mL of water, but to delay all morning-time medication (apart from metformin) until conclusion of the examination day. After taking subjects history, current weight and blood pressure, intravenous catheters will be placed in both forearms after which blood and urine will be collected. Thereupon the combined renal and clamp protocol will commence.

Safety and tolerability: Telephone consultation and follow-up Participants will be asked about the occurrence of adverse events and the intake of study drugs will be checked. Furthermore, recent history will be taken, physical examination/anthropometric measurements performed and blood and urine samples collected.

Study Procedures Renal protocol During this protocol a combined inulin/para-aminohippurate (PAH)-clearance technique will be performed to examine the glomerular filtration rate (GFR, ml/min) and effective renal plasma flow (ERPF, ml/min) respectively. In order to examine tubular function, sodium, potassium, chloride, calcium, magnesium, phosphate, urea and glucose will be measured in urine (mmol). In addition, urine osmolality will be determined. Moreover, biomarkers of renal damage (urinary albumin excretion (UAE), Neutrophil gelatinase-associated lipocalin (NGAL) and Kidney Injury Molecule-1 (KIM-1) will be measured in urine

Clamp protocol A combined hyperinsulinemic-euglycemic and hyperglycemic clamp will be performed. During the euglycemic clamp insulin will be infused at 40 microunits/square meter.minute (mU/m2.min) and glucose will be kept at 5 mmol/l by variable glucose 20% infusion. This technique allows for renal measurements during normoglycemia in all participants. After 3 hours of insulin infusion and an one hour rest period for exogenous insulin to be cleared, glucose will be infused in order to reach a plasma concentration of 15 mmol/l. In this matter, renal tests can be performed under stable hyperglycemia. From the euglycemic clamp, insulin sensitivity will be determined from the amount of glucose infused (M-value). Blood will be stored during hyperglycemia in order to be able to obtain measures of beta-cell function, including 1st phase insulin secretion, 2nd phase insulin secretion and arginine-induced insulin secretion.

(cardio)vascular measures After an acclimatization period of >5 minutes, blood pressure will be measured three times at the non-dominant arm, with an automatic oscillometric device (Dinamap®, General Electric (GE) Healthcare). Systemic hemodynamics will be measured by an automated, beat-to-beat blood pressure and ECG recording monitor (Nexfin®, BMEYE, Amsterdam, The Netherlands). Body composition will be assessed by bio impedance analysis using tetrapolar Soft Tissue Analyzer® (STA, Akern, Florence, Italy). Microvascular function will be measured by nail fold skin capillary density on the middle finger, and skin blood flow will be measured using a Laser Doppler probe. Applanation tonometry using the SphygmoCor® system (Atcor Medical, West Ryde, Australia) will be performed to measure variables of arterial stiffness at the radial artery of the non-dominant arm.

Fecal examinations Each participant will collect a stool sample before the baseline tests and once before the long-term follow-up tests. At home, one feces sample must be stored at room temperature and one in the freezer and when arrived at the CRU, the feces will be stored at -20⁰C and -80⁰C, respectively.

SAFETY (REPORTING) In accordance with the guidelines of ICH-GCP, the European Clinical Trials Directive (2001/20/EC) and the local regulations, the investigator will inform the subjects and the reviewing Ethical Review Board (ERB) if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal.

Reporting The investigator will be responsible for reporting the SAEs and SUSARs to the accredited ERB. This will be done within 15 days after first knowledge, using the specified web portal ('ToetsingOnline'), which automatically leads to informing the respective national health authorities. For fatal or life threatening SAEs and SUSARs this term will be 7 days for a preliminary report ('expedited') with another 8 days for completion of the report.

The involved pharmaceutical company (AstraZeneca) will be notified of all SAEs, pregnancy, clinical relevant overdosing and adverse events of special interest (AESIs), if any.

Monitoring As required by GCP, a monitoring procedure will be performed in order to oversee the progress of the clinical trial and ensure that it is conducted, recorded and reported in accordance with the protocol, standard operating procedures (SOPs), GCP and the applicable regulatory requirements.

Statistical Analysis Plan All tests of differences between treatments will be conducted at a two-sided significance level of <0.05. In case of missing data, a multiple imputation technique will be applied and compared with complete case analysis. The efficacy analysis population will be based on the per protocol (PP) principle - i.e. all subjects who completed the entire treatment period using the treatment as originally allocated. Safety analysis will be performed in all patients who received one or more doses of the study medication.

In order to compare the effects between the two study arms the investigators will perform t-tests and/or multivariable linear regression models. The latter technique allows us to use continuous outcome variables and both continuous and dichotomous independent variables. The efficacy endpoint of interest will be added to the model as dependent variable.

Our primary outcomes will be the most important outcomes for testing the hypothesis that SGLT-2 inhibitor dapagliflozin versus the SU gliclazide causes an improvement in renal hemodynamics. The large amount of secondary/exploratory endpoints potentially justifies the use of corrections for multiple tests. However, there is an increasing debate on whether this should be done, because of the increased risk of type 2 errors which could lead to prematurely discarding of potential useful observations. As recently pointed out, in a hypothesis-generating study - such as the current study - correction for multiple outcomes can be detrimental. A final decision will be made in the detailed Statistical Analysis Plan (SAP) prior to the conduction of the analysis.

13. ETHICS The trial will be conducted in accordance with the Declaration of Helsinki (64th World Medical Association (WMA) General Assembly, Fortaleza, Brazil, October 2013) for biomedical research involving human subjects and in accordance with ICH-GCP. The investigator will ensure that all aspects of the institutional ERB review are conducted in accordance with current institutional, local and national regulations.

Study Medication Participants will be randomized for a 12 week treatment with two different active study agents. Consequently, independent of treatment allocation, beneficial effects can be expected, as both SGLT-2 inhibitors and SU derivatives improve glycemic control. Both study medications have been approved for blood-glucose lowering treatment in T2DM patients and, based on currently available data, are considered to be safe. Furthermore, SGLT-2 inhibitors in general may decrease blood pressure and body weight compared to gliclazide.

The most common side effects for dapagliflozin are hypoglycemia (especially when used in combination with a SU derivative or insulin) and genital mycotic- and urinary tract infections. For gliclazide, hypoglycemia and blurred vision in the initiation phase of treatment (due to changes in blood glucose levels) are the most common side effects. As in all drug intervention trials, in this study, the investigators will closely monitor patients for adverse drug and study events during the follow-up visit and by telephone consultation according to GCP. Participants can contact the research staff 24 hours a day.

Safety issues The study examinations/tests are considered to be safe. No invasive procedures (besides intravenous peripheral catheters) are involved. During the study tests, two 'diagnostic agents' (i.e. inulin and PAH) need to be administered; both agents are inert and have no side effects. The total amount of drawn blood will be 500 mL during a total period of 16 weeks. Side effects are not expected because the blood volume taken per visit is relatively small, especially in comparison with regular blood donation, with 500 mL per donation (and is allowed 5 times a year for men and 3 times for women).

Publication policy AstraZeneca will be provided will all intended publication(s) and abstract(s), preceding submission at least 30 days and 7 days, respectively, AstraZeneca can make suggestions to change the wording of any planned publication or abstract in relation to the study and/or the results. The sponsor-investigator is under no obligation to implement such changes, unless local regulatory requirements specify otherwise.

Data will be presented at relevant national and international scientific meetings, and published in peer reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian*
* Both genders (females must be post-menopausal; no menses >1 year; in case of doubt, Follicle-Stimulating Hormone (FSH) will be determined with cut-off defined as >31 U/L)
* Age: 35 - 75 years
* BMI: >25 kg/m2
* HbA1c: 6.5 - 9.0% Diabetes Control and Complications Trial (DCCT) or 48 - 86 mmol/mol International Federation of Clinical Chemistry (IFCC)
* Treatment with a stable dose of oral antihyperglycemic agents for at least 3 months prior to inclusion
* Metformin monotherapy
* Combination of metformin and low dose SU derivative**
* Hypertension should be controlled, i.e. ≤140/90 mmHg, and treated with an ACE-I or ARB (unless prevented by side effect) for at least 3 months.
* Albuminuria should be treated with a RAAS-interfering agent (ACE-I or ARB) for at least 3 months.
* Written informed consent

  * In order to increase homogeneity ** In order to accelerate inclusion, patients using combined metformin/SU derivative will be considered. In these patients, a 12 week wash-out period of the SU derivative will be observed, only when combined use has led to a HbA1c <8% at screening. Subsequently, patients will be eligible to enter the study, now using metformin monotherapy, provided that HbA1c still meets inclusion criteria.

Exclusion Criteria:

* History of unstable or rapidly progressing renal disease
* Macroalbuminuria; defined as albumin-creatinine ratio of 300mg/g.
* Estimated GFR <60 mL/min/1.73m2 (determined by the Modification of Diet in Renal Disease (MDRD) study equation)
* Current/chronic use of the following medication: thiazolidinedione (TZD), SU derivative, Glucagon like peptide 1 receptor agonist (GLP-1RA), (dipeptidyl peptidase 4 inhibitor) DPP-4I, SGLT-2 inhibitors, glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors (MAOIs). Subjects on diuretics will only be excluded when these drugs cannot be stopped for the duration of the study.
* Volume depleted patients. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status.
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, head-ache or back ache). However, no such drugs can be taken within a time-frame of 2 weeks prior to renal-testing
* History of diabetic ketoacidosis (DKA) requiring medical intervention (eg, emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including:

  * Acute coronary syndrome
  * Chronic heart failure (New York Heart Association grade II-IV)
  * Stroke or transient ischemic neurologic disorder
* Complaints compatible with neurogenic bladder and/or incomplete bladder emptying (as determined by ultrasonic bladder scan)
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* (Unstable) thyroid disease; defined as free thyroxine (fT4) outside of laboratory reference values or change in treatment within 3 months prior to screening visit
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day)
* Allergy to any of the agents used in the study
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study
* Inability to understand the study protocol or give informed consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-02; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark HH Kramer, MD/PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Suijk DLS, van Baar MJB, van Bommel EJM, Iqbal Z, Krebber MM, Vallon V, Touw D, Hoorn EJ, Nieuwdorp M, Kramer MMH, Joles JA, Bjornstad P, van Raalte DH. SGLT2 Inhibition and Uric Acid Excretion in Patients with Type 2 Diabetes and Normal Kidney Function. Clin J Am Soc Nephrol. 2022 May;17(5):663-671. doi: 10.2215/CJN.11480821. Epub 2022 Mar 23. PMID 35322793
- [Derived] van Baar MJB, van Bommel EJM, Smits MM, Touw DJ, Nieuwdorp M, Ten Kate RW, Joles JA, van Raalte DH. Whole-body insulin clearance in people with type 2 diabetes and normal kidney function: Relationship with glomerular filtration rate, renal plasma flow, and insulin sensitivity. J Diabetes Complications. 2022 Apr;36(4):108166. doi: 10.1016/j.jdiacomp.2022.108166. Epub 2022 Feb 20. PMID 35221224
- [Derived] van Bommel EJM, Geurts F, Muskiet MHA, Post A, Bakker SJL, Danser AHJ, Touw DJ, van Berkel M, Kramer MHH, Nieuwdorp M, Ferrannini E, Joles JA, Hoorn EJ, van Raalte DH. SGLT2 inhibition versus sulfonylurea treatment effects on electrolyte and acid-base balance: secondary analysis of a clinical trial reaching glycemic equipoise: Tubular effects of SGLT2 inhibition in Type 2 diabetes. Clin Sci (Lond). 2020 Dec 11;134(23):3107-3118. doi: 10.1042/CS20201274. PMID 33205810
- [Derived] van Bommel EJM, Smits MM, Ruiter D, Muskiet MHA, Kramer MHH, Nieuwdorp M, Touw DJ, Heerspink HJL, Joles JA, van Raalte DH. Effects of dapagliflozin and gliclazide on the cardiorenal axis in people with type 2 diabetes. J Hypertens. 2020 Sep;38(9):1811-1819. doi: 10.1097/HJH.0000000000002480. PMID 32516291
- [Derived] van Bommel EJM, Lytvyn Y, Perkins BA, Soleymanlou N, Fagan NM, Koitka-Weber A, Joles JA, Cherney DZI, van Raalte DH. Renal hemodynamic effects of sodium-glucose cotransporter 2 inhibitors in hyperfiltering people with type 1 diabetes and people with type 2 diabetes and normal kidney function. Kidney Int. 2020 Apr;97(4):631-635. doi: 10.1016/j.kint.2019.12.021. No abstract available. PMID 32200854
- [Derived] van Bommel EJM, Herrema H, Davids M, Kramer MHH, Nieuwdorp M, van Raalte DH. Effects of 12-week treatment with dapagliflozin and gliclazide on faecal microbiome: Results of a double-blind randomized trial in patients with type 2 diabetes. Diabetes Metab. 2020 Apr;46(2):164-168. doi: 10.1016/j.diabet.2019.11.005. Epub 2019 Dec 6. PMID 31816432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Started | 24 | 20
Completed | 24 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7) | 63 (7) | 63 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 19 | 15 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate (GFR) in ml/Min
Description: Calculated from urinary and plasma inulin concentrations, GFR in ml/min
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
ml/min | 104 (17) | 109 (20)

2. Primary Outcome: Effective Renal Plasma Flow (ERPF) in ml/Min
Description: Calculated from urinary and plasma para-aminohippurate concentrations, ERPF in ml/min
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
ml/min | 639 (141) | 678 (122)

3. Secondary Outcome: Fractional Excretion of Sodium in % of Filtered Sodium
Description: Calculated fractional excretions with measured GFR (see above) and urinary and plasma concentrations of sodium. Fractional excretion in % of filtered sodium
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of filtered sodium
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
% of filtered sodium | 0.74 (0.19) | 0.66 (0.22)

4. Secondary Outcome: Fractional Excretion of Potassium in % of Filtered Potassium
Description: Calculated fractional excretions with measured GFR (see above) and urinary and plasma concentrations of potassium. Fractional excretion in % of filtered potassium
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of filtered potassium
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
% of filtered potassium | 13.6 (3.3) | 11.8 (3.4)

5. Secondary Outcome: Fractional Excretion of Glucose in % of Filtered Glucose
Description: Calculated fractional excretions with measured GFR (see above) and urinary and plasma concentrations of glucose. Fractional excretion in % of filtered glucose
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of filtered glucose
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
% of filtered glucose | 31.1 (15.6) | 0.6 (1)

6. Secondary Outcome: Urinary Albumin-Creatinine Ratio in mg/mmol
Description: Calculated from measured urinary albumin and creatinin concentrations, in mg/mmol
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/mmol
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
mg/mmol | 0.88 [0.31 to 1.48] | 0.54 [0.31 to 1.30]

7. Secondary Outcome: Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: NGAL (ng/mmoll) measured in urine as a marker of renal damage
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mmol
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
ng/mmol | 3.76 [2.24 to 5.84] | 3.79 [2.80 to 6.29]

8. Secondary Outcome: Kidney Injury Molecule-1 (KIM-1) in ng/mmol
Description: KIM-1 (ng/mmol) measured in urine as a marker of renal damage
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mmol
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
ng/mmol | 0.25 [0.105 to 0.288] | 0.265 [0.160 to 0.548]

9. Other Pre Specified Outcome: Body Weight
Description: Measured in kilograms
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
kilograms | 93.7 (16.9) | 99.6 (18.3)

10. Other Pre Specified Outcome: Systolic Blood Pressure
Description: Blood pressure will be measured using an automated oscillometric blood pressure device (Dinamap®) in mmHg
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
Number analyzed (Participants) | 24 | 20
mmHg | 129.2 (10.7) | 131.1 (11.8)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Dapagliflozin 10mg Once Daily | Gliclazide Modified Release 30mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 5/24 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg Once Daily (N=24) | Gliclazide Modified Release 30mg Once Daily (N=20)
genital fungal infections (Renal and urinary disorders) | 5 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
For GFR measurements, iohexol was used instead of inulin because inulin was retracted for human use during the trial. This did not alter our findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02682563/Prot_SAP_000.pdf